CLINICAL TRIAL: NCT02425930
Title: The Relationship Between Complement C3 Depletion and Metastatic Gastric Cancer: A Prospective Pilot Study
Brief Title: The Predictive Value of Complement C3 in Patients With Advanced Gastric Cancer
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yulong He, Director of Center of Gastrointestinal Surgery, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: [2013]A-246
Record Dates: First submitted 2015-04-10; First posted 2015-04-24 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Gastric Cancer; Complement Component Deficiency; Surgery
Keywords: gastric cancer; complement system; overal survival
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gastrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- C3 Depletion: Patients with persistent low-level of complement C3 within the perioperative period would be assigned into this main observational group. After a careful multidisciplinary treatment (MDT) discussion, a radical operation with gastrectomy plus D2 lymphadenectomy would be performed, followed by an adjuvant chemotherapy if required. Generally, SOX chemo regimen (S-1+Oxaliplatin) would be first considered for the candidates.
  Interventions: Procedure: gastrectomy plus D2 lymphadenectomy; Drug: S-1+Oxaliplatin
- Non-C3 depletion: Patients with normal plasma values of complement C3 within the perioperative period would be assigned into this control group. Those patients would undergo the same decision making process to determine the final treatment plan.
  Interventions: Procedure: gastrectomy plus D2 lymphadenectomy; Drug: S-1+Oxaliplatin

INTERVENTIONS:
Procedure: gastrectomy plus D2 lymphadenectomy — A classic total or subtotal gastrectomy plus D2 lymph nodes dissection would be performed for all enrolled patients. Patients in both groups would undergo the identical therapeutic approach for gastric cancer, mainly decided by a multidisciplinary treatment group in our center.
  Other Names: D2 surgery
Drug: S-1+Oxaliplatin — A postoperative systemic chemotherapy would be performed for some subjects who have advanced gastric cancer. The concrete chemo regimen for adjuvant chemotherapy is also determined by a MDT group. Generally, SOX chemo regimen is the first-line treatment in our center, as following described:
  * S-1: 40~60mg bid，po, Day1~14 （S-1：BSA <1.25m2, 40mg bid, 1.25m2≤BSA≤1.5m2,50mg bid, BSA>1.5m2, 60mg bid）
  * Oxaliplatin: 130mg/m2，iv drip for 2h，Day1
  Other Names: SOX regimen

SUMMARY:
This study is designed to investigate whether complement C3 depletion is associated with poor short-term outcomes in postoperative patients with gastric cancer.

DETAILED DESCRIPTION:
The complement system plays an important role in the development of digestive malignancies. The complement C3 is the point of convergence for the three complement activation pathways. However, the concrete effect of C3 in the development of gastric cancer is still obscured. This study is designed to explore whether complement C3 can be regarded as a predictive factor of postoperative outcomes for postoperative patients with gastric cancer.

This study is designed as a prospective cohort study and included consecutively treated patients. The perioperative plasma value of complement components, such as C3, C4, and CH50, are detected to explore the incidence rate of complement depletion. All enrolled patients are divided into two groups mainly according to the levels of preoperative C3 levels (C3 depletion and Non-C3 depletion groups). The primary endpoints are the 1-year overall survival and disease-free survival, while the secondary endpoints are postoperative complications, length of hospital stay, and hospital charges.

This study would be helpful to confirm the role of complement depletion in anticipated outcomes of postoperative patients with gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathological diagnosis of gastric adenocarcinoma
* Radical operation and adjuvant chemotherapy endurable
* Informed consent approved

Exclusion Criteria:

* Age <18 or >75 years old
* Pregnancy or lactating woman
* Any primary diagnosis other than gastric cancer
* Confirmed complement deficiency due to immunity dysfunction or other disease
* Required blood transfusion, plasmapheresis, or emergent operation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have a confirmed pathological diagnosis of gastric adenocarcinoma would be selected for further observation. Those patients who subsequently underwent a radical tumor resection can be included for final analysis.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2013-08; Primary Completion 2015-02 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Overall Survival | one year after surgery
  1-year overall survival (OS) would be regarded as primary endpoint of this study.
Disease-Free Survival | One year after surgery
  1-year disease-free survival (DFS) would be also regarded as primary endpoint of this study.

SECONDARY OUTCOMES:
Early complications | within 30 days after a radical operation
  Early postoperative events should include intra-abdominal infection, postoperative hemorrhage, anastomotic leak, surgical site infection, ileus, and so on. Number of such events would be recorded to calculate incidence.
Length of hospital stay | an expected average of 4 weeks after admission
  Time frame would cover the period from admission to discharge from hospital. An average of 4 weeks is expected.
Expenditure of hospitalization | an expected average of 4 weeks after admission
  The total costs during the hospitalization would be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Yulong He, MD, Principal Investigator — First Hospital, Sun Yat-sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Yuan K, Ye J, Liu Z, Ren Y, He W, Xu J, He Y, Yuan Y. Complement C3 overexpression activates JAK2/STAT3 pathway and correlates with gastric cancer progression. J Exp Clin Cancer Res. 2020 Jan 13;39(1):9. doi: 10.1186/s13046-019-1514-3. PMID 31928530